CLINICAL TRIAL: NCT00703053
Title: A Phase II Randomized Study of the Safety and Immunogenicity of Vaccination Strategies Using One or Two Clades and Different Schedules of H5N1 Unadjuvanted, Inactivated Subvirion Influenza Vaccines in H5 Naïve Healthy Adults
Brief Title: H5N1 Priming and Boosting Strategies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-0019; N01AI80003C
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2009-09

CONDITIONS: Influenza
Keywords: influenza, H5N1, vaccine, avian influenza, parent protocol
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- Group 1 (Experimental): 25 subjects: Day 0, A/Vietnam/04 90 mcg; Day 7, A/Vietnam/04 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04
- Group 9 (Experimental): 100 subjects: Day 0, A/Vietnam/04 90 mcg; Day 28, A/Vietnam/04 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04
- Group 8 (Experimental): 100 subjects: Day 0, A/Vietnam/04 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04
- Group 7 (Experimental): 50 subjects: Day 0, A/Indonesia/05 90 mcg; Day 180, A/Indonesia/05 90 mcg.
  Interventions: Biological: A/Indonesia/05/05
- Group 6 (Experimental): 50 subjects: Day 0, A/Vietnam/04 90 mcg; Day 180, A/Indonesia/05 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04; Biological: A/Indonesia/05/05
- Group 5 (Experimental): 50 subjects: Day 0, A/Vietnam/04 45 mcg + A/Indonesia/05 45 mcg; Day 28, A/Vietnam/04 45 mcg + A/Indonesia/05 45 mcg.
  Interventions: Biological: A/Vietnam/1203/04; Biological: A/Indonesia/05/05
- Group 4 (Experimental): 50 subjects: Day 0, A/Vietnam/04 90 mcg; Day 28, A/Indonesia/05 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04; Biological: A/Indonesia/05/05
- Group 3 (Experimental): 50 subjects: Day 0, A/Indonesia/05 90 mcg; Day 28, A/Indonesia/05 90 mcg.
  Interventions: Biological: A/Indonesia/05/05
- Group 2 (Experimental): 25 subjects: Day 0, A/Vietnam/04 90 mcg; Day 14, A/Vietnam/04 90 mcg.
  Interventions: Biological: A/Vietnam/1203/04

INTERVENTIONS:
Biological: A/Vietnam/1203/04 — Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine; dosages 45 mcg and 90 mcg.
  Arms: Group 1; Group 2; Group 4; Group 5; Group 6; Group 8; Group 9
Biological: A/Indonesia/05/05 — Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine; dosages 45 mcg and 90 mcg.
  Arms: Group 3; Group 4; Group 5; Group 6; Group 7

SUMMARY:
Severe disease in humans due to bird influenza viruses (H5N1) has led to concern that this virus may result in a widespread outbreak of bird flu. The purpose of this study is to evaluate the dose and dosing schedule for 2 different types of H5N1 vaccine. Participants will be randomly assigned to 1 of 9 possible vaccine groups. All participants will receive 2 doses of Clade 1, Clade 2, or combination Clade 1 and 2 on Day 0. All participants will receive a second dose of the same vaccine or a different vaccine type on study day 7, 14, 28 or 180. Study participants will include about 500 healthy adult subjects, ages 18-49 years old, who have no history of prior H5 flu exposure or vaccination. Study procedures may include medical history, physical exam, and blood sampling. Subject participation may last up to 372 days. Several DMID studies have recently evaluated H5N1 vaccines in healthy adults, 04-063, 05-0090, 05-0015, and 05-0043.

DETAILED DESCRIPTION:
Severe disease in humans due to avian influenza viruses of the H5N1 subtype has raised concern regarding the potential emergence of these viruses in pandemic form. Results of earlier studies suggest that previous priming can significantly affect the responses to subsequent booster doses, even if these booster doses represent an antigenic variant. Both the length of time between priming and revaccination, as well as the antigenic relatedness of the priming and revaccination antigens, may impact the response. These issues could have an important impact on pre-vaccination strategies prior to the emergence of a pandemic. This study will evaluate immunogenicity with the same or with different H5 variants. In this study, "different" will be defined as clade 1 followed by clade 1, clade 1 followed by clade 2, clade 2 followed by clade 2, or a combination of clades 1 & 2 followed by a combination of clades 1 & 2. In addition, the study will evaluate the effect of the interval between doses on the subsequent response, with "ultra-short" intervals defined as 7 or 14 days, a "short" interval defined as 28 days and a "long" interval defined as 180 days. The study will evaluate whether the use of a longer duration between doses or cross-clade priming will result in enhanced immunogenicity. Primary objectives are: evaluate the dose and schedules of unadjuvanted inactivated subvirion H5N1 vaccines belonging to the same or different clades in H5-naïve, healthy adults; determine if boosting of subjects given the inactivated influenza rg A/Vietnam/1203/04 vaccine with a heterologous antigen inactivated influenza rg A/Indonesia/05/05 results in broader or higher immune responses compared with boosting with the homologous antigen; and evaluate the immune response to 2 doses of H5 vaccine given at times < 1 month apart. Secondary objectives are: determine the safety of 2 doses of inactivated H5 vaccines in healthy adults given at different schedules and antigen combinations; obtain additional information regarding the antibody response to a single dose and to ultra-short immunization schedules; and evaluate the effect on antibody levels after receiving an antigenic variant to the priming virus given as a booster or simultaneously. The study will be conducted as a randomized, prospective controlled, multi-center trial. Approximately 500 healthy adult subjects, aged 18-49, who have no history of prior H5 influenza exposure or vaccination will be enrolled. Subjects will be randomized to receive varying schedules, (2 doses separated by 7, 14, 28 or 180 days), and clades of unadjuvanted inactivated subvirion H5N1 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 through 49 years old, who deny exposure to H5 virus or participation in an H5 vaccine study.
* In good health, as determined by vital signs (heart rate less than 100 bpm; blood pressure: systolic less than or equal to 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature less than 100.0 degrees Fahrenheit), medical history to ensure stable medical condition and a targeted physical examination, as indicated, based on medical history. A stable medical condition is defined as no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to 1 year) must not be pregnant as indicated by a negative pregnancy test (urine or serum) within 24 hours prior to vaccine administration.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier methods, abstinence, monogamous relationship with vasectomized partner, intrauterine devices, Depo-Provera, Norplant, oral contraceptives, contraceptive patches or other licensed, effective methods) until 30 days following receipt of the last dose of vaccine.
* Able to understand and comply with planned study procedures.
* Able to provide informed consent prior to initiation of any study procedures and be available for all study visits.

Exclusion Criteria:

* Has occupational exposure to poultry, to include but is not limited to chicken, turkey, or duck farmer, factory worker in poultry processing plant, veterinary staff that handles poultry; has recreational exposure to poultry, e.g. raising poultry in 4-H club, duck hunter that slaughters/handles the "kill" or history of previous H5N1 vaccination or exposure.
* Has a known allergy to eggs, egg products or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal and egg or chicken protein).
* Is female of child-bearing potential who is breastfeeding or intends to become pregnant during the study period up to 30 days following receipt of the last dose of vaccine.
* Has immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. Active neoplastic disease is defined as no neoplastic disease or treatment for neoplastic disease within the past 5 years.
* Has long-term use (greater than 2 weeks) of oral or parenteral steroids (glucocorticoids), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood products within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study, or plans to receive any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) following each study vaccine.
* Has an acute or chronic medical condition that would render vaccination unsafe or would interfere with the evaluation of responses. This includes, but is not limited to solicited reactogenicity symptoms, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.
* Has a history of severe reactions following vaccination with contemporary influenza virus vaccines.
* Has an acute illness or has an oral temperature greater than 99.9 degrees Fahrenheit (37.7 degrees Celsius) within 3 days prior to enrollment.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the study period.
* Has any condition that would, in the opinion of the site principal investigator place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has a diagnosis of schizophrenia, bipolar disease or other severe (disabling) chronic psychiatric diagnosis.
* Has been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Is receiving psychiatric drugs. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Has known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Has a history of alcohol or drug abuse in the 5 years prior to enrollment.
* Has a history of Guillain-Barré syndrome.
* Has any condition that the investigator believes may interfere with successful completion of the study.
* Plans to enroll in another clinical trial (that has a study intervention in the form of drug, biologic or device that could interfere with safety assessment of H5N1 vaccine) at any time during the study period.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 505 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia
  - Mayo Clinic, Rochester - Vaccine Research Group, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Group Health Cooperative, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Belshe RB, Frey SE, Graham I, Mulligan MJ, Edupuganti S, Jackson LA, Wald A, Poland G, Jacobson R, Keyserling HL, Spearman P, Hill H, Wolff M; National Institute of Allergy and Infectious Diseases-Funded Vaccine and Treatment Evaluation Units. Safety and immunogenicity of influenza A H5 subunit vaccines: effect of vaccine schedule and antigenic variant. J Infect Dis. 2011 Mar 1;203(5):666-73. doi: 10.1093/infdis/jiq093. Epub 2011 Jan 31. PMID 21282194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy ambulatory adults were recruited from the surrounding communities of the research clinics from September 8, 2008 to November 12, 2008.
Groups:
- VN/VN, Day 0, 7: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage; Day 7, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage.
- VN/VN, Day 0, 14: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage; Day 14, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage.
- I/I, Day 0, 28: Day 0, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage; Day 28, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage.
- VN/I, Day 0, 28: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage; Day 28, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage.
- VN+I/VN+I, Day 0, 28: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 45 mcg dosage and Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 45 mcg dosage; Day 28, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 45 mcg dosage and Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 45 mcg dosage.
- VN/I, Day 0, 180: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage; Day 180, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage.
- I/I, Day 0, 180: Day 0, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage; Day 180, Inactivated subvirion influenza rg A/Indonesia/05/05 (clade 2) x PR8 A/H5N1 vaccine (I); 90 mcg dosage.
- VN, Day 0: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage.
- VN/VN, Day 0, 28: Day 0, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage; Day 28, Inactivated subvirion influenza rg A/Vietnam/1203/04 (clade 1) x PR8 A/H5N1 vaccine (VN); 90 mcg dosage.
Period: Overall Study
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Started | 27 | 26 | 51 | 49 | 51 | 49 | 52 | 97 | 103
Completed | 26 | 24 | 48 | 46 | 50 | 43 | 45 | 91 | 102
Not Completed | 1 | 2 | 3 | 3 | 1 | 6 | 7 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28 | Total
Number analyzed (Participants) | 27 | 26 | 51 | 49 | 51 | 49 | 52 | 97 | 103 | 505
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 51 | 49 | 51 | 49 | 52 | 97 | 103 | 505
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.6 (9.6) | 34.0 (9.5) | 37.0 (9.2) | 33.6 (7.9) | 31.9 (8.8) | 33.8 (9.3) | 33.5 (9.6) | 34.3 (9.4) | 35.2 (8.4) | 34.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 36 | 31 | 24 | 26 | 30 | 60 | 61 | 296
  Male | 13 | 12 | 15 | 18 | 27 | 23 | 22 | 37 | 42 | 209
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 51 | 49 | 51 | 49 | 52 | 97 | 103 | 505

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) Against A/Vietnam/04 Antigen
Description: The GMTs are as assessed by the HAI assay against the A/Vietnam/04 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: Analyses are based on a modified intent to treat population. 1 subject is excluded at all timepoints due to steroid receipt. 21 subjects not receiving vaccination 2 and one misdosed at vaccination 2 were dropped at timepoints post vaccination 2 only, as were 5 due to receipt of prohibited vaccines/steroids.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Titer | 14.7 [7.6 to 28.5] | 27.9 [11.6 to 67.0] | 6.7 [5.2 to 8.7] | 13.6 [8.8 to 20.9] | 15.1 [9.4 to 24.1] | 39.7 [23.7 to 66.4] | 10.5 [7.7 to 14.1] | 9.1 [7.0 to 11.6] | 22.9 [16.3 to 32.2]

2. Secondary Outcome: Number of Serious Adverse Events
Description: Serious adverse events were collected at each study visit from the time of first vaccination through the final study visit at 180 days after the last vaccination.
Time Frame: Duration of study
Population: All subjects receiving at least one study vaccination are included in the safety population and analyses of safety are intention to treat (ITT). Three subjects were randomized but not vaccinated.
Measure: Number; unit: Events
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 25 | 51 | 48 | 51 | 49 | 52 | 97 | 103
Events | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms Within 7 Days of First Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after first vaccination and review the Memory Aid with clinic staff at follow a up visit on Day 8. Subjects are counted if they indicated experiencing the symptom at any severity during the reporting period. The symptoms of redness and swelling were solicited as both functional grading as impact on daily activies as well as collected as a measured value in mm. The number reported for all symptoms is the number reporting greater than none.
Time Frame: 7 days after first vaccination
Population: All subjects receiving the first vaccination are included in the safety population and analyses of safety are ITT. Three subjects were randomized but not vaccinated.
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 25 | 51 | 48 | 51 | 49 | 52 | 97 | 103
Participants
  Fever | 1 | 1 | 2 | 3 | 4 | 1 | 3 | 5 | 9
  Malaise | 2 | 4 | 10 | 13 | 16 | 9 | 11 | 25 | 28
  Myalgia | 5 | 8 | 13 | 12 | 13 | 9 | 12 | 23 | 25
  Headache | 5 | 11 | 19 | 18 | 20 | 15 | 14 | 32 | 40
  Nausea | 2 | 1 | 2 | 5 | 5 | 2 | 3 | 9 | 11
  Pain | 9 | 11 | 10 | 14 | 20 | 28 | 15 | 38 | 44
  Tenderness | 17 | 15 | 21 | 35 | 27 | 30 | 20 | 66 | 76
  Redness (functional) | 3 | 6 | 6 | 7 | 10 | 7 | 6 | 7 | 15
  Redness (measured) | 3 | 6 | 12 | 9 | 16 | 10 | 8 | 13 | 19
  Swelling (functional) | 0 | 3 | 3 | 2 | 5 | 5 | 2 | 5 | 11
  Swelling (measured) | 1 | 4 | 4 | 3 | 6 | 5 | 3 | 6 | 12

4. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms Within 7 Days of Second Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after the second vaccination and review the Memory Aid with clinic staff at a follow up visit on Day 8. Subjects are counted if they indicated experiencing the symptom at any severity during the reporting period. The symptoms of redness and swelling were solicited as both functional grading as impact on daily activies as well as collected as a measured value in mm. The number reported for all symptoms is the number reporting greater than none.
Time Frame: 7 days after second vaccination
Population: All subjects receiving the second vaccination are included in this outcome measure. The VN, Day 0 Group received only one dose.
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 46 | 44 | 48 | 45 | 47 | 97
Participants
  Fever | 0 | 2 | 3 | 1 | 5 | 3 | 3 | 6
  Malaise | 3 | 4 | 8 | 4 | 13 | 6 | 9 | 24
  Myalgia | 5 | 4 | 5 | 5 | 12 | 5 | 5 | 22
  Headache | 7 | 8 | 8 | 11 | 12 | 10 | 13 | 22
  Nausea | 4 | 2 | 3 | 2 | 2 | 2 | 5 | 11
  Pain | 9 | 8 | 12 | 7 | 19 | 10 | 11 | 49
  Tenderness | 15 | 14 | 21 | 24 | 28 | 26 | 22 | 71
  Redness (functional) | 4 | 2 | 7 | 3 | 3 | 7 | 7 | 11
  Redness (measured) | 7 | 4 | 11 | 5 | 7 | 10 | 8 | 22
  Swelling (functional) | 1 | 2 | 5 | 1 | 2 | 5 | 2 | 9
  Swelling (measured) | 3 | 3 | 6 | 1 | 4 | 6 | 3 | 13

5. Secondary Outcome: Neutralizing Geometric Mean Titer (GMT) Against A/Vietnam/04 Antigen
Description: The GMTs are as assessed by the microneutralization assay against the A/Vietnam/04 antigen at 1 month following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Titer | 9.1 [6.6 to 12.6] | 12.6 [7.5 to 21.2] | 5.8 [5.1 to 6.5] | 9.8 [7.5 to 12.6] | 9.6 [7.7 to 11.9] | 56.6 [37.2 to 86.0] | 10.9 [8.6 to 13.9] | 7.1 [6.1 to 8.3] | 17.0 [13.7 to 21.0]

6. Secondary Outcome: Neutralizing Geometric Mean Titer (GMT) Against A/Indonesia/05 Antigen
Description: The GMTs are as assessed by the microneutralization assay against the A/Indonesia/05 antigen at 1 month following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Titer | 5.3 [5.0 to 5.7] | 6.1 [5.4 to 6.9] | 70.0 [49.0 to 100.0] | 21.5 [15.7 to 29.4] | 66.8 [46.2 to 96.5] | 85.3 [54.4 to 133.8] | 183.2 [127.1 to 264.2] | 5.4 [5.1 to 5.7] | 7.2 [6.5 to 7.9]

7. Secondary Outcome: Number of Subjects Achieving a 4-fold or Greater Neutralizing Antibody Titer Increase Against A/Vietnam/04 Antigen
Description: The number of subjects who achieve a 4-fold or greater rise in titer, relative to the baseline (Day 0) titer, assessed by the microneutralization assay against the A/Vietnam/04 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations. Subjects whose baseline titer is <10 must have a post vaccination titer of at least 1:40 to be considered a 4-fold rise.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 3 | 6 | 1 | 7 | 3 | 28 | 6 | 7 | 30

8. Primary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) Against A/Indonesia/05 Antigen
Description: The GMTs are as assessed by the HAI assay against the A/Indonesia/05 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Titer | 5.1 [4.9 to 5.2] | 5.1 [4.9 to 5.2] | 27.6 [16.8 to 45.5] | 10.1 [7.1 to 14.4] | 24.3 [15.1 to 39.2] | 41.3 [22.9 to 74.7] | 58.7 [38.0 to 90.7] | 5.3 [4.8 to 5.9] | 5.7 [5.2 to 6.3]

9. Primary Outcome: Number of Subjects Achieving a 4-fold or Greater HAI Antibody Titer Increase Against A/Vietnam/04 Antigen
Description: The number of subjects who achieve a 4-fold or greater rise in titer, relative to the baseline (Day 0) titer, assessed by the HAI assay against the A/Vietnam/04 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations. Subjects whose baseline titer is <10 must have a post vaccination titer of at least 1:40 to be considered a 4-fold rise.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 8 | 10 | 3 | 11 | 14 | 25 | 8 | 14 | 41

10. Primary Outcome: Number of Subjects Achieving a 4-fold or Greater HAI Antibody Titer Increase Against A/Indonesia/05 Antigen
Description: The number of subjects who achieve a 4-fold or greater rise in titer, relative to the baseline (Day 0) titer, assessed by the HAI assay against the A/Indonesia/05 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations. Subjects whose baseline titer is <10 must have a post vaccination titer of at least 1:40 to be considered a 4-fold rise.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 0 | 0 | 23 | 9 | 22 | 24 | 32 | 1 | 3

11. Primary Outcome: Number of Subjects Achieving a HAI Antibody Titer of 1:40 or Greater Against A/Vietnam/04 Antigen
Description: The number of subjects who achieve a HAI antibody titer of 1:40 or greater as assessed by the HAI assay against the A/Vietnam/04 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 8 | 10 | 3 | 11 | 14 | 25 | 8 | 14 | 41

12. Primary Outcome: Number of Subjects Achieving a HAI Antibody Titer of 1:40 or Greater Against A/Indonesia/05 Antigen
Description: The number of subjects who achieve a HAI antibody titer of 1:40 or greater as assessed by the HAI assay against the A/Indonesia/05 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 0 | 0 | 23 | 9 | 22 | 24 | 32 | 1 | 3

13. Secondary Outcome: Number of Subjects Achieving a 4-fold or Greater Neutralizing Antibody Titer Increase Against A/Indonesia/05 Antigen
Description: The number of subjects who achieve a 4-fold or greater rise in titer, relative to the baseline (Day 0) titer, assessed by the microneutralization assay against the A/Indonesia/05 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations. Subjects whose baseline titer is <10 must have a post vaccination titer of at least 1:40 to be considered a 4-fold rise.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 0 | 0 | 34 | 14 | 34 | 30 | 43 | 1 | 1

14. Secondary Outcome: Number of Subjects Achieving Neutralizing Antibody Titer of 1:40 or Greater Against A/Vietnam/04 Antigen
Description: The number of subjects who achieve a titer of 1:40 or greater as assessed by the microneutralization assay against the A/Vietnam/04 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 3 | 6 | 1 | 7 | 3 | 28 | 6 | 7 | 30

15. Secondary Outcome: Number of Subjects Achieving Neutralizing Antibody Titer of 1:40 or Greater Against A/Indonesia/05 Antigen
Description: The number of subjects who achieve a titer of 1:40 or greater as assessed by the microneutralization assay against the A/Indonesia/05 antigen at 28 days following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: 28 days post last vaccination.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 45 | 43 | 48 | 43 | 46 | 94 | 95
Participants | 0 | 0 | 34 | 14 | 34 | 30 | 43 | 1 | 1

16. Secondary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) Against A/Vietnam/04 Antigen at 6 Months Post Last Vaccination
Description: The GMTs are as assessed by the HAI assay against the A/Vietnam/04 antigen at 6 months following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: Six months post last vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 25 | 23 | 44 | 41 | 47 | 42 | 44 | 91 | 95
Titer | 8.8 [5.3 to 14.6] | 9.0 [5.1 to 15.9] | 6.1 [4.9 to 7.8] | 6.6 [5.2 to 8.2] | 7.7 [5.5 to 10.7] | 8.3 [5.9 to 11.6] | 5.5 [4.7 to 6.4] | 7.3 [5.8 to 9.0] | 10.4 [8.2 to 13.1]

17. Secondary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) Against A/Indonesia/05 Antigen at 6 Months Post Last Vaccination
Description: The GMTs are as assessed by the HAI assay against the A/Indonesia/05 antigen at 6 months following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations. The CI shown as 5.0 to 5.0 reflect that all subjects had a titer of 5.0 for the VN,VN, Day 0,14 and VN, Day 0 groups.
Time Frame: Six months after last vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 25 | 23 | 44 | 41 | 47 | 42 | 44 | 91 | 95
Titer | 5.4 [4.6 to 6.5] | 5.0 [5.0 to 5.0] | 7.8 [5.7 to 10.6] | 6.4 [5.1 to 8.0] | 6.2 [5.2 to 7.4] | 6.7 [5.2 to 8.6] | 8.4 [6.2 to 11.4] | 5.0 [5.0 to 5.0] | 5.2 [5.0 to 5.4]

18. Secondary Outcome: Neutralizing Geometric Mean Titer (GMT) Against A/Vietnam/04 Antigen at 6 Months Post Last Vaccination
Description: The GMTs are as assessed by the microneutralization assay against the A/Vietnam/04 antigen at 6 months following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: Six months post last vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 25 | 23 | 44 | 41 | 47 | 42 | 44 | 91 | 95
Titer | 5.8 [4.6 to 7.4] | 8.3 [5.7 to 12.3] | 5.3 [4.9 to 5.7] | 6.2 [5.3 to 7.4] | 6.4 [5.6 to 7.4] | 7.7 [6.3 to 9.3] | 5.2 [4.9 to 5.4] | 5.8 [5.3 to 6.3] | 8.5 [7.4 to 9.8]

19. Secondary Outcome: Neutralizing Geometric Mean Titer (GMT) Against A/Indonesia/05 Antigen at 6 Months Post Last Vaccination
Description: The GMTs are as assessed by the microneutralization assay against the A/Indonesia/05 antigen at 6 months following the last vaccination. One group (VN, Day 0) receives only one vaccination, all other groups receive two vaccinations.
Time Frame: Six months post last vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Number analyzed (Participants) | 25 | 23 | 44 | 41 | 47 | 42 | 44 | 91 | 95
Titer | 5.5 [4.9 to 6.2] | 6.0 [5.2 to 7.0] | 20.6 [15.8 to 26.9] | 16.1 [11.7 to 22.1] | 18.4 [14.0 to 24.1] | 14.7 [11.8 to 18.4] | 23.0 [18.2 to 29.2] | 5.5 [5.2 to 5.7] | 5.9 [5.5 to 6.4]

20. Secondary Outcome: Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) Against A/Vietnam/04 Antigen at 1, 2, 3 and 4 Weeks After 2 Doses
Description: The kinetics of the antibody response to vaccination with A/Vietnam/04 is evaluated by the HAI GMT against the A/Vietnam/04 antigen at weekly intervals after receipt of 2 doses 7, 14 and 28 days apart
Time Frame: Weeks 1, 2, 3 and 4 after the second dose
Population: Analyses are based on a modified intent to treat population. 5 subjects in the VN/VN, Day 0, 28 group not receiving vaccination 2 are excluded, as were 2, also in this group, due to receipt of prohibited vaccines.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | VN/VN, Day 0, 28
Number analyzed (Participants) | 26 | 24 | 95
Titer
  Week 1 | 16.2 [8.0 to 32.8] | 33.2 [14.2 to 77.6] | 23.5 [16.6 to 33.2]
  Week 2 | 18.5 [8.8 to 38.8] | 32.4 [12.7 to 82.4] | 29.9 [20.7 to 43.2]
  Week 3 | 16.2 [7.8 to 33.3] | 28.7 [11.9 to 69.4] | 30.9 [22.1 to 43.3]
  Week 4 | 14.7 [7.6 to 28.5] | 27.9 [11.6 to 67.0] | 22.9 [16.3 to 32.2]

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected for 7 days after each vaccination, unsolicited non-serious adverse events were collected through 28 days after each vaccination. Serious adverse events were collected through 180 days after the last vaccination.
Description: For the solicited symptoms, subjects are counted if reporting the symptom after either vaccination, with the occurrence within 0-7 days of a vaccination considered 1 event.
Arm/Group | VN/VN, Day 0, 7 | VN/VN, Day 0, 14 | I/I, Day 0, 28 | VN/I, Day 0, 28 | VN+I/VN+I, Day 0, 28 | VN/I, Day 0, 180 | I/I, Day 0, 180 | VN, Day 0 | VN/VN, Day 0, 28
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/25 | 0/51 | 0/48 | 0/51 | 0/49 | 1/52 | 0/97 | 0/103
Other Adverse Events (participants affected / at risk) | 23/26 | 23/25 | 44/51 | 42/48 | 42/51 | 46/49 | 39/52 | 85/97 | 98/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VN/VN, Day 0, 7 (N=26) | VN/VN, Day 0, 14 (N=25) | I/I, Day 0, 28 (N=51) | VN/I, Day 0, 28 (N=48) | VN+I/VN+I, Day 0, 28 (N=51) | VN/I, Day 0, 180 (N=49) | I/I, Day 0, 180 (N=52) | VN, Day 0 (N=97) | VN/VN, Day 0, 28 (N=103)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VN/VN, Day 0, 7 (N=26) | VN/VN, Day 0, 14 (N=25) | I/I, Day 0, 28 (N=51) | VN/I, Day 0, 28 (N=48) | VN+I/VN+I, Day 0, 28 (N=51) | VN/I, Day 0, 180 (N=49) | I/I, Day 0, 180 (N=52) | VN, Day 0 (N=97) | VN/VN, Day 0, 28 (N=103)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (4)
Reactogenicity event (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 8 (8) | 7 (9) | 7 (7) | 6 (6) | 3 (3) | 9 (9) | 26 (26)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 5 (5) | 3 (4) | 8 (9) | 4 (4) | 6 (6) | 5 (5) | 12 (15) — Oral temperature was measured daily for days 0-7 after vaccination. Temperatures 37.8 degrees Celsius or greater were considered fever.
Malaise (General disorders) | 4 (5) | 5 (8) | 16 (18) | 14 (17) | 19 (29) | 12 (15) | 15 (20) | 25 (25) | 39 (52) — Solicited for Days 0-7 after each vaccination as "Fatigue/Malaise (feeling unwell)" on the Memory Aid.
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 9 (12) | 17 (18) | 14 (17) | 18 (25) | 11 (14) | 16 (17) | 23 (23) | 36 (47) — Solicited for Days 0-7 after each vaccination as "Myalgia(Muscle aches/pains)" on the Memory Aid.
Headache (Nervous system disorders) | 9 (12) | 13 (19) | 21 (27) | 23 (29) | 24 (32) | 20 (25) | 19 (27) | 32 (32) | 48 (62) — Solicited for Days 0-7 after each vaccination as "Headache" on the Memory Aid.
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (3) | 5 (5) | 7 (7) | 7 (7) | 4 (4) | 7 (8) | 9 (9) | 20 (22) — Solicited for Days 0-7 after each vaccination as "Nausea" on the Memory Aid.
Injection site pain (General disorders) | 11 (18) | 13 (19) | 17 (22) | 18 (21) | 23 (39) | 31 (38) | 20 (26) | 38 (38) | 65 (93) — Solicited for Days 0-7 after each vaccination as "Pain" under Injection Site Reactions on the Memory Aid.
Tenderness (General disorders) | 18 (32) | 18 (29) | 29 (42) | 37 (59) | 34 (55) | 36 (56) | 29 (42) | 66 (66) | 90 (147) — Solicited for Days 0-7 after each vaccination as "Tenderness" under Injection Site Reactions on the Memory Aid.
Injection site erythema (functional grading) (General disorders) | 5 (7) | 7 (8) | 11 (13) | 7 (10) | 11 (13) | 10 (14) | 11 (13) | 7 (7) | 18 (26) — Solicited for Days 0-7 after each vaccination as "Erythema/Redness" under Injection Site Reactions on the Memory Aid.
Injection site erythema (measured values) (General disorders) | 8 (10) | 8 (10) | 20 (23) | 11 (14) | 19 (23) | 14 (20) | 12 (16) | 13 (13) | 28 (41) — Solicited for Days 0-7 after each vaccination as "Erythema/Redness" under Injection Site Reactions on the Memory Aid. Subjects measured the diameter of observed erythema. Measurements greater than 0 are counted as the reaction occurring.
Injection site swelling (functional grading) (General disorders) | 1 (1) | 4 (5) | 6 (8) | 3 (3) | 7 (7) | 8 (10) | 3 (4) | 5 (5) | 15 (20) — Solicited for Days 0-7 after each vaccination as "Induration/Swelling" under Injection Site Reactions on the Memory Aid on a scale of impact on daily activities.
Injection site swelling (measured values) (General disorders) | 4 (4) | 5 (7) | 8 (10) | 4 (4) | 9 (10) | 9 (11) | 4 (6) | 6 (6) | 20 (25) — Solicited for Days 0-7 after each vaccination as "Induration/Swelling" under Injection Site Reactions on the Memory Aid. Subjects measured the diameter of observed swelling. Measurements greater than 0 are counted as the reaction occurring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less